CLINICAL TRIAL: NCT03600428
Title: Clinical Study of the Safety of Quadrivalent Live Attenuated Influenza Vaccine (LAIV4) in Children With Asthma of Varying Levels of Severity
Brief Title: Safety of LAIV4 in Children With Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Duke University (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Buddy Creech, Associate Professor of Pediatrics, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 181211; 200-2012-50430 Task Order 0005 (Other Grant/Funding Number: Centers for Disease Control and Prevention)
Record Dates: First submitted 2018-07-11; First posted 2018-07-26 (Actual); Results first posted 2021-02-25 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-02

CONDITIONS: Asthma in Children; Vaccine Adverse Reaction; Vaccine Reaction; Asthma; Wheezing; Influenza
Keywords: asthma; influenza vaccine; inactivated influenza vaccine; live attenuated influenza vaccine
MeSH Terms: conditions — Asthma; Respiratory Sounds; Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Live Attenuated Influenza Vaccine (LAIV) (Experimental): Participants will receive one dose of live attenuated influenza vaccine via intranasal spray (administer approximately one half of the contents of the single-dose intranasal sprayer into each nostril, each sprayer contains 0.2 mL of vaccine)).
  Interventions: Biological: Live Attenuated Influenza Vaccine (LAIV)
- Inactivated Influenza Vaccine (IIV) (Active Comparator): Participants will receive one dose of inactivated influenza vaccine via intramuscular injection (0.5 mL).
  Interventions: Biological: Inactivated Influenza Vaccine (IIV)

INTERVENTIONS:
Biological: Live Attenuated Influenza Vaccine (LAIV) — 1 dose, 0.2 mL, intranasal administration
  Arms: Live Attenuated Influenza Vaccine (LAIV)
Biological: Inactivated Influenza Vaccine (IIV) — 1 dose, 0.5 mL, intramuscular administration
  Arms: Inactivated Influenza Vaccine (IIV)

SUMMARY:
This is a prospective randomized, open label clinical trial in approximately 300 children aged 5-11 years with a physician diagnosis of persistent asthma. Participants will be randomized 1:1 to receive either a single intranasal dose of licensed quadrivalent LAIV (LAIV4) or an intramuscular injection of quadrivalent IIV4 (IIV4).

DETAILED DESCRIPTION:
The study will be conducted at three sites: Vanderbilt University Medical Center (Lead site), Cincinnati Children's Hospital Medical Center (contributing site), and Duke University Medical Center (contributing site) during the 2018-2019 influenza season. Participants will be randomized 1:1 to receive either a single intranasal dose of licensed quadrivalent LAIV (LAIV4) or an intramuscular injection of quadrivalent IIV4 (IIV4), stratifying by asthma severity (mild vs. moderate-to-severe). Vanderbilt will enroll about 100 participants, Cincinnati will enroll about 110 participants, and Duke will enroll about 90 participants. After enrollment, participants will be followed for 43 days via 5 additional phone, email, or text visits to monitor systemic reactogenicity, asthma symptoms and exacerbations, and serious adverse events. The primary objective is to compare proportions of participants with asthma exacerbations during the 42 days after LAIV4 versus IIV4. Because of the potential for increased risk of wheezing after LAIV, the use of LAIV in persons with asthma has been an area of vaccine safety research for many years; the safety issue remains unresolved. A clinical study to assess the safety of LAIV4 in children with asthma could expand the evidence base and inform clinical decision-making and public health policy.

ELIGIBILITY:
Inclusion Criteria:

* Children between 5-11 years of age, inclusive, at enrollment
* Participant must have a current diagnosis of persistent asthma (Physician diagnosis of asthma and current prescribed use of a long-acting controller medication. For purposes of this study, we have considered "controller" medications to be any single or combination use of long-acting medications used to prevent asthma exacerbations and to achieve long-term control of asthma (as compared to short-acting rescue medication).)
* Parent(s) or legal guardian(s) must provide written, informed consent and participant must provide assent as appropriate for age prior to initiation of study procedures and according to local IRB requirements
* Parent(s) or legal guardian(s) and participant must be willing and able to comply with planned study procedures and be available for all study visits
* Is in good health, other than their asthma, as determined by medical history
* English or Spanish literate (only English-speaking participants will be included at the Cincinnati and Duke sites)
* Intention of being available for entire study period and complete all relevant study procedures, including follow-up using at least one of the following methods: phone calls, text messages, or emails

Exclusion Criteria:

* Acute illness and/or a reported oral temperature of ≥ 100.4°F within 72 hours prior to enrollment (this may result in a temporary delay of vaccination)
* Use of antipyretic medication during the preceding 24 hours that might mask a fever (this may result in a temporary delay of vaccination)
* History of a severe allergic reaction (e.g., anaphylaxis) after a previous dose of any influenza vaccine or after any component of the influenza vaccine, including egg protein.
* Receipt of any licensed vaccine within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to vaccination or planned receipt of any licensed vaccine within 42 days after vaccination
* Receipt of current year's (2018-2019 influenza season) licensed influenza vaccine for children 9-11 years (only). (Clarification: Children aged 5-8 years are permitted to be enrolled if they have received zero or one dose of the 2018-2019 influenza season vaccine, and require two doses of the 2018-2019 influenza vaccine.)
* Received an investigational agent (licensed or unlicensed vaccine, drug, biologic, device, blood product, or medication) in the 28 days prior to enrollment or planned receipt before 42 days after vaccination
* Have immunosuppression as a result of an underlying illness or treatment, or use of anticancer chemotherapy or radiation therapy within the preceding 36 months
* Have taken ≥20mg/day of prednisone or its equivalent, for 14 days or more within the past 28 days
* Have known active neoplasm or a history of any hematologic malignancy
* Has had a previous exacerbation of their asthma symptoms requiring systemic steroids within the prior 28 days, or has had a life-threatening exacerbation of asthma in the past two years (e.g. hypoxic seizure, mechanical ventilation)
* Received influenza antiviral medication within 48 hours prior to study vaccination
* History of Guillian-Barré syndrome within 6 weeks of previous influenza vaccination
* Have any condition that, in the opinion of the investigator, would interfere with the evaluation of the responses or would place the participant at unacceptable risk of injury
* Has a positive urine or serum pregnancy test within 24 hours prior to vaccination in a post-menarchal female. LAIV is not recommended for use in pregnant females.
* Currently taking aspirin or aspirin-containing products
* Any parent(s) or legal guardian(s) who is an immediate relative of study staff or is an employee supervised by study staff.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 152 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Buddy Creech, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (3):
- United States (3):
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sokolow AG, Stallings AP, Kercsmar C, Harrington T, Jimenez-Truque N, Zhu Y, Sokolow K, Moody MA, Schlaudecker EP, Walter EB, Staat MA, Broder KR, Creech CB. Safety of Live Attenuated Influenza Vaccine in Children With Asthma. Pediatrics. 2022 Apr 1;149(4):e2021055432. doi: 10.1542/peds.2021-055432. PMID 35342923

RESULTS

PARTICIPANT FLOW:
Groups:
- Live Attenuated Influenza Vaccine (LAIV4): Participants will receive one dose of quadrivalent live attenuated influenza vaccine via intranasal spray (administer approximately one half of the contents of the single-dose intranasal sprayer into each nostril, each sprayer contains 0.2 mL of vaccine)).
  Quadrivalent Live Attenuated Influenza Vaccine (LAIV4): 1 dose, 0.2 mL, intranasal administration
- Inactivated Influenza Vaccine (IIV4): Participants will receive one dose of quadrivalent inactivated influenza vaccine via intramuscular injection (0.5 mL).
  Quadrivalent Inactivated Influenza Vaccine (IIV4): 1 dose, 0.5 mL, intramuscular administration
Period: Overall Study
Arm/Group | Live Attenuated Influenza Vaccine (LAIV4) | Inactivated Influenza Vaccine (IIV4)
Started | 79 | 73
15-day Follow-up | 76 | 70
43-day Follow-up | 74 | 68
Completed | 74 | 68
Not Completed | 5 | 5
Not completed — Not eligible | 0 | 1
Not completed — Lost to Follow-up | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Live Attenuated Influenza Vaccine (LAIV4) | Inactivated Influenza Vaccine (IIV4) | Total
Number analyzed (Participants) | 79 | 72 | 151
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 9.00 [7.00 to 12.00] | 9.00 [7.00 to 11.00] | 9.00 [7.00 to 12.00]
Age, Customized [Count of Participants; unit: Participants]
  Age Group: 5-11 years old | 58 | 55 | 113
  Age Group: 12-17 years old | 21 | 17 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 28 | 63
  Male | 44 | 44 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 75 | 69 | 144
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 24 | 49
  White | 43 | 42 | 85
  More than one race | 9 | 6 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race recoded: White | 43 | 42 | 85
  Race recoded: Black | 25 | 24 | 49
  Race recoded: Other | 11 | 6 | 17
Site [Count of Participants; unit: Participants]
  Vanderbilt | 12 | 8 | 20
  Cincinnati | 54 | 53 | 107
  Duke | 13 | 11 | 24
Asthma Severity Status [Count of Participants; unit: Participants]
  Mild | 26 | 19 | 45
  Moderate or Severe | 53 | 53 | 106
Weight in kg [Median (Inter-Quartile Range); unit: kilograms] | 39.1 [27.4 to 50.0] | 35.0 [24.9 to 52.6] | 38.3 [25.7 to 51.4]
Height [Median (Inter-Quartile Range); unit: inches] | 53.90 [49.65 to 60.10] | 53.70 [49.21 to 60.95] | 53.75 [49.46 to 60.15]
BMI [Median (Inter-Quartile Range); unit: kg/m2] | 19.50 [16.45 to 22.90] | 18.60 [16.15 to 21.65] | 18.75 [16.30 to 22.50]
Received seasonal influenza vaccine in the past 12 months [Count of Participants; unit: Participants]
  No | 42 | 43 | 85
  Yes | 30 | 26 | 56
  Unknown | 7 | 3 | 10
History of nasal or sinus allergies [Count of Participants; unit: Participants]
  No | 19 | 27 | 46
  Yes | 56 | 45 | 101
  Unknown | 4 | 0 | 4
Influenza Season [Count of Participants; unit: Participants]
  2018-2019 | 27 | 25 | 52
  2019-2020 | 52 | 47 | 99

OUTCOME MEASURES:

1. Primary Outcome: Comparison of the Proportion of Participants Experiencing an Asthma Exacerbation During the 42 Days After LAIV4 vs. IIV4 (Until Day 43).
Description: For this study, asthma exacerbation will be defined as: any acute episode of progressively worsening shortness of breath (dyspnea), cough, wheezing, chest tightness, and/or respiratory distress during the 42 days (until day 43) after influenza vaccination for which the patient seeks unscheduled medical attention (e.g., healthcare provider office or Emergency Department visit or hospitalization) or receives a new prescription for systemic corticosteroids.
Time Frame: Day 43
Measure: Count of Participants; unit: Participants
Groups:
- Live Attenuated Influenza Vaccine (LAIV4): Participants received one dose of quadrivalent live attenuated influenza vaccine via intranasal spray (administer approximately one half of the contents of the single-dose intranasal sprayer into each nostril, each sprayer contains 0.2 mL of vaccine)).
  Quadrivalent Live Attenuated Influenza Vaccine (LAIV4): 1 dose, 0.2 mL, intranasal administration
- Inactivated Influenza Vaccine (IIV4): Participants received one dose of quadrivalent inactivated influenza vaccine via intramuscular injection (0.5 mL).
  Quadrivalent Inactivated Influenza Vaccine (IIV4): 1 dose, 0.5 mL, intramuscular administration
Arm/Group | Live Attenuated Influenza Vaccine (LAIV4) | Inactivated Influenza Vaccine (IIV4)
Number analyzed (Participants) | 74 | 68
Participants
  Asthma exacerbation within 43 days | 8 | 10
  No asthma exacerbation within 43 days | 66 | 58

2. Secondary Outcome: Comparison of the Proportion of Participants Experiencing an Asthma Exacerbation During the 14 Days After LAIV4 vs. IIV4
Description: For this study, asthma exacerbation will be defined as: any acute episode of progressively worsening shortness of breath (dyspnea), cough, wheezing, chest tightness, and/or respiratory distress during the 14 days (until day 15) after influenza vaccination for which the patient seeks unscheduled medical attention (e.g., healthcare provider office or Emergency Department visit or hospitalization) or receives a new prescription for systemic corticosteroids.
Time Frame: Day 15
Measure: Count of Participants; unit: Participants
Arm/Group | Live Attenuated Influenza Vaccine (LAIV4) | Inactivated Influenza Vaccine (IIV4)
Number analyzed (Participants) | 76 | 70
Participants
  Asthma exacerbation within 14 days | 3 | 4
  No asthma exacerbation within 14 days | 73 | 66

3. Secondary Outcome: Comparison of the Proportion of Participants With Asthma Symptoms and Unscheduled Albuterol Use During the 14 Days After Receipt of LAIV4 or IIV4 (Each is Assessed Separately).
Description: Cough, wheezing, tightness in chest, nighttime awakening and unscheduled albuterol use will all be assessed by parent self-report
Time Frame: Day 15
Measure: Count of Participants; unit: Participants
Arm/Group | Live Attenuated Influenza Vaccine (LAIV4) | Inactivated Influenza Vaccine (IIV4)
Number analyzed (Participants) | 76 | 70
Participants
  Asthma symptoms within 14 days: No | 18 | 20
  Asthma symptoms within 14 days: Yes | 58 | 50
  Night-time awakening within 14 days: No | 55 | 42
  Night-time awakening within 14 days: Yes | 21 | 28
  Unscheduled Albuterol use within 14 days: No | 41 | 44
  Unscheduled Albuterol use within 14 days: Yes | 35 | 26

4. Secondary Outcome: Comparison of the Proportion of Participants With Asthma Symptoms and Unscheduled Albuterol Use During the 14 Days After Receipt of LAIV4 or IIV4 (Each is Assessed Separately).
Description: as for outcome 3
Time Frame: Day 15
Measure: Count of Participants; unit: Participants
Arm/Group | Live Attenuated Influenza Vaccine (LAIV4) | Inactivated Influenza Vaccine (IIV4)
Number analyzed (Participants) | 76 | 70
Participants
  Asthma related cough within 14 days: None | 26 | 22
  Asthma related cough within 14 days: Mild | 35 | 29
  Asthma related cough within 14 days: Moderate | 14 | 15
  Asthma related cough within 14 days: Severe | 1 | 4
  Asthma related wheezing within 14 days: None | 51 | 39
  Asthma related wheezing within 14 days: Mild | 19 | 18
  Asthma related wheezing within 14 days: Moderate | 5 | 12
  Asthma related wheezing within 14 days: Severe | 1 | 1
  Asthma related chest tightness within 14 days: None | 58 | 45
  Asthma related chest tightness within 14 days: Mild | 12 | 21
  Asthma related chest tightness within 14 days: Moderate | 5 | 3
  Asthma related chest tightness within 14 days: Severe | 1 | 1

5. Secondary Outcome: Comparison of the Proportion of Participants Who Experience a Clinically Significant Decrease in Peak Flow Measurement From Baseline During the 14 Days After LAIV4 or IIV4
Description: For purposes of this measure, a clinically significant decrease in peak flow is defined as: a decrease of ≥20% in PEFR from baseline PEFR
Time Frame: Baseline, Day 15
Measure: Count of Participants; unit: Participants
Arm/Group | Live Attenuated Influenza Vaccine (LAIV4) | Inactivated Influenza Vaccine (IIV4)
Number analyzed (Participants) | 76 | 70
Participants
  No PEFR decrease >= 20% from baseline within 14 days | 36 | 37
  PEFR decreased >= 20% from baseline within 14 days | 39 | 33
  Unknown | 1 | 0

ADVERSE EVENTS:
Time Frame: Within 42 days (until day 43) after vaccination.
Description: Adverse events (AEs), including serious adverse events (SAEs) were recorded on the memory aid and included the need for new prescription or nonprescription medications for the control of asthma, an unscheduled healthcare provider visit or consultation, any other clinically significant event at any point during the study period. The definition of SAEs matched the definition from clinicaltrials.gov.
Arm/Group | Live Attenuated Influenza Vaccine (LAIV4) | Inactivated Influenza Vaccine (IIV4)
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/68
Other Adverse Events (participants affected / at risk) | 8/74 | 10/68
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Live Attenuated Influenza Vaccine (LAIV4) (N=74) | Inactivated Influenza Vaccine (IIV4) (N=68)
Asthma Exacerbation (Respiratory, thoracic and mediastinal disorders) | 8 | 10 — Any acute episode of progressively worsening shortness of breath, cough, wheezing, chest tightness, and/or respiratory distress for which the patient seeks unscheduled medical attention or receives a new prescription for systemic corticosteroids.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-07-03): https://cdn.clinicaltrials.gov/large-docs/28/NCT03600428/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/28/NCT03600428/SAP_001.pdf